CLINICAL TRIAL: NCT04737070
Title: Study of High Risk Non Invasive Prenatal Test Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Matthieu DAP, medical doctor (MD), Central Hospital, Nancy, France
Other Study IDs: 2020PI310
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Trisomy 21
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Prenatal test for Trisomy 21 screening — prenatal routine test for Trisomy 21 screening (blood test + nuchal translucency test)

SUMMARY:
The investigator want to study the population of high risk (over 1/50) of Trisomy 21.

According to french guidelines, these patients needs to have a invasive test (such as amniocentesis) but some patients prefer to have a Non Invasive Prenatal Test, with a potential lack of information.

ELIGIBILITY:
Inclusion Criteria:

* Prenatal screening of Trisomy 21 > 1/50 (high risk population)

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High risk population for prenatal screening of Trisomy 21
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
number of genetics anomalies | through study completion, an average of 9 months

IPD SHARING:
Plan to Share IPD: Undecided